CLINICAL TRIAL: NCT04091035
Title: Prevalence and Risk Factors for Common Diseases in Sweden: A Nationwide Cohort Study
Brief Title: Prevalence and Risk Factors for Common Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Anna Nordström (Other Government)
Collaborators: Umeå University (Other)
Responsible Party: Sponsor-Investigator, Anna Nordström, Associate professor, Region Västerbotten
Organization: Region Västerbotten (Other Government)
Other Study IDs: VasterbottenCounty
Record Dates: First submitted 2019-09-13; First posted 2019-09-16 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Cardiovascular Diseases; Fracture; Cancer
MeSH Terms: conditions — Cardiovascular Diseases; Fractures, Bone; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: To describe the incidence of disease and evaluate risk factors — Se above

SUMMARY:
By using national databases in Sweden the aim of the present project is to:

1. Investigate if the incidence of our most common diseases, such as fracture and cardiovascular disease, has changed from 1970-2017
2. To investigate whether the risk of death for our most common diseases have changed from 1970-2017.
3. To investigate the risk of a new episode after suffering from our most common diseases from 1970-2017
4. To investigate the risk factors for our most common diseases, and whether these have changed from 1970.
5. To investigate how severe disease or death affects the health of a close relative.

DETAILED DESCRIPTION:
Please see above on the summary.

ELIGIBILITY:
Inclusion Criteria:

* All people living in Sweden that is diagnosed with our most common diseases between 1970-2017.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Se above
Sampling Method: Non-Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of disease | 1970-2017
  To investigate the incidence of the most common diseases, and whether the incidence has changed.
Age at diagnosis of disease | 1970-2017
  To investigate age at diagnosis of our most common diseases, and whether this has changed.
Risk of death or disease in relative | 1970-2017
  Risk of death or disease in close relative to those diagnosed with severe disease or died.
Risk factors for disease or death | 1970-2017
  Risk factors for our most common diseases or death

SECONDARY OUTCOMES:
Risk for readmission | 1970-2017
  To investigate the risk of readmission for our most common diseases, and whether this risk has changed,

CONTACTS AND LOCATIONS:
Overall Officials: Peter Nordström, Professor, Study Director — Umea University

IPD SHARING:
Plan to Share IPD: No